CLINICAL TRIAL: NCT00470015
Title: Melanoma Peptide Vaccines (MART1 Analog, gp100 and Survivin) With GM-CSF and Low-Dose IL-2 as Immune Adjuvants, A Pilot Study
Brief Title: Vaccine Therapy and GM-CSF With or Without Low-Dose Aldesleukin in Treating Patients With Stage II, Stage III, or Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000542631; P30CA015083 (NIH); MC0575 (Other: Mayo Clinic Cancer Center); 06-002650 (Other: Mayo Clinic IRB); NCI-2009-1306 (Registry Identifier: NCI-CTRP)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; Interleukin-2; aldesleukin; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MART1 Analog, gp100 and Survivin (Experimental)
  Interventions: Biological: MART-1 antigen; Biological: IL-2; Biological: gp100 antigen; Biological: GM-CSF; Biological: MART-1a peptide

INTERVENTIONS:
Biological: MART-1 antigen — 1000 mcg; Day 1 of a 21 day cycle x 4
Biological: IL-2 — 0.5x10^6/m^2
  Other Names: Interleukin-2, Proleukin®, aldesleukin
Biological: gp100 antigen — 1000 mcg; Day 1 of a 21 day cycle x 4
Biological: GM-CSF — 300mcg
  Other Names: Leukine-Liquid, sargramostatin
Biological: MART-1a peptide — 1000 mcg; Day 1 of a 21 day cycle x 4

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Aldesleukin may stimulate the white blood cells to kill tumor cells. Giving vaccine and different doses of GM-CSF mixed in incomplete Freund's adjuvant, with or without aldesleukin, may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and how well giving vaccine therapy together with GM-CSF, with or without low-dose aldesleukin, works in treating patients with stage II, stage III, or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity profile of peptide vaccine comprising MART-1 antigen, gp100 antigen, and survivin antigen in combination with sargramostim (GM-CSF) emulsified in incomplete Freund's adjuvant (IFA) with or without low-dose aldesleukin in patients with stage II-IV melanoma.
* Determine the immunologic effects of two different doses of GM-CSF coemulsified with melanoma peptides in IFA in these patients.
* Determine the immunological effects of low-dose aldesleukin therapy administered after peptide immunization in these patients.
* Collect preliminary data on the impact of the vaccine on clinical outcomes in these patients.

OUTLINE: This is a pilot study. Patients are stratified according to disease stage (II vs III or IV). Patients are sequentially enrolled into 1 of 4 different dose schedules.

* Dose schedule 1: Patients receive gp100 antigen, MART-1 antigen, survivin antigen, and sargramostim (GM-CSF) emulsified in incomplete Freund's adjuvant (peptide vaccine) subcutaneously (SC) on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Dose schedule 2: Patients receive peptide vaccine as in group 1. Patients also receive low-dose aldesleukin SC twice daily on days 7-20. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Dose schedule 3: Patients receive peptide vaccine as in group 1 except with a higher dose of GM-CSF. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Dose schedule 4: Patients receive peptide vaccine as in group 1 except with a higher dose of GM-CSF. Patients also receive low-dose aldesleukin SC twice daily on days 7-20. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 5 patients receive treatment at subsequent dose schedule until the maximum tolerated dose schedule (MTDS) is determined. The MTDS is defined as the dose schedule preceding that at which 2 of 5 patients experience dose-limiting toxicity within the first course.

After completion of study therapy, patients are followed every 3 months for up to 2 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma

  * Stage II-IV disease
* Completely resected disease
* No known standard therapy that is potentially curative or proven capable of extending life expectancy exists
* HLA-A2 positive

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm³
* Hemoglobin > 10 g/dL
* Platelet count ≥ 50,000/mm³
* AST ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled or current infection
* No known allergy to vaccine or immunoadjuvant components
* No known immune deficiency

PRIOR CONCURRENT THERAPY:

* No chemotherapy within the past 4 weeks and recovered
* No biologic therapy within the past 4 weeks
* No radiation therapy within the past 4 weeks

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-03 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2013-01-02 (Actual)

PRIMARY OUTCOMES:
Percent changes in peptide vaccine-specific immune responses (tetramer frequencies) from pretreatment levels | 12 weeks
Number and severity of hematologic and nonhematologic toxicities observed at each dose level | 12 weeks

SECONDARY OUTCOMES:
Delayed-type hypersensitivity positivity | 12 weeks
Maximum percent change in CD4, CD8, CD14, CD19, and C20 levels from preimmunization levels | 12 weeks
Time to treatment failure | 12 weeks
Time to progression | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, MD, PhD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States